CLINICAL TRIAL: NCT02072343
Title: The Effect of 10 cm Catheter Mount on Malfunction of Capnometers Under the Conditions of Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Wonhee Kim, Emergency medicine fellow, Hanyang University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Capnometry with DCCM
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Cardiopulmonary Resuscitation; Pulmonary Edema; Hemorrhage
Keywords: Capnography; Catheters; Intubation
MeSH Terms: conditions — Pulmonary Edema; Hemorrhage | interventions — Water

ARMS (2):
- Mainstream capnometer (Experimental)
  Interventions: Device: No-DCCM; Device: DCCM; Other: Water 5ml in tracheal tube; Other: Water 10ml in tracheal tube
- Microstream capnograph (Experimental)
  Interventions: Device: No-DCCM; Device: DCCM; Other: Water 5ml in tracheal tube; Other: Water 10ml in tracheal tube

INTERVENTIONS:
Device: No-DCCM
  Other Names: Proximal capnometer of DCCM; Abbreviation: DCCM, direct connect catheter mount
Device: DCCM
  Other Names: Distal capnometer of DCCM; Abbreviation: DCCM, direct connect catheter mount
Other: Water 5ml in tracheal tube
Other: Water 10ml in tracheal tube

SUMMARY:
Capnometer has been used to assess the success of intubation and the quality of cardiopulmonary resuscitation. However, capnometers can malfunction under the conditions such as pulmonary edema and hemorrhage due to the vulnerability of capnometers for water. Investigators hypothesized that the use of 10cm catheter mount will reduce the malfunction of capnometers under the conditions of water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults without underlying disease

Exclusion Criteria:

* Lung and heart disease
* Drinking carbonated beverages

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
the malfunction rate of capnograph | 1 day
  The malfunction of capnograph is defined that the ETCO2 level is out-of the measured range of each patient under water-free conditions. The calculation formula of malfunction rate is as follows: malfunctioning time of capnograph / total experiment time (2min).
  1. Water conditions in tracheal tube
     * Water 5ml
     * Water 10ml
  2. Capnometers
     * Mainstream capnometer
     * Microstream capnograph
  3. Comparison group
     * No-DCCM group (proximal capnometer of DCCM)
     * DCCM group (distal capnometer of DCCM)
  Abbreviation : DCCM, Direct connect catheter mount

SECONDARY OUTCOMES:
The cumulative survival rate of capnometers under the conditions of water | 1 day
  1. Kaplan-Meier analysis
  1-1. Water conditions in tracheal tube
  * Water 5ml
  * Water 10ml
  1-2. Capnometers
  * Mainstream capnometer
  * Microstream capnograph
  1-3. Comparison group
  * No-DCCM group (proximal capnometer of DCCM)
  * DCCM group (distal capnometer of DCCM)
  Abbreviation : DCCM, Direct connect catheter mount
The consistency of ETCO2 between No-DCCM group and DCCM group under the water-free conditions | 1 day
  1. Bland-Altman plots under water 0ml in tracheal tube.
     1-1. Capnometers
     * Mainstream capnometer
     * Microstream capnograph
     1-3. Comparison group
     * No-DCCM group (proximal capnometer of DCCM)
     * DCCM group (distal capnometer of DCCM)
  2. The intraclass correlation coefficient (ICC) under water 0ml in tracheal tube
  2-1. Capnometers
  * Mainstream capnometer
  * Microstream capnograph
  2-2. Comparison group
  * No-DCCM group (proximal capnometer of DCCM)
  * DCCM group (distal capnometer of DCCM)

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University, Seoul, South Korea